CLINICAL TRIAL: NCT01526499
Title: Docetaxel With or Without Metronomic Cyclophosphamide as First Line Chemotherapy in Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, yanfei Liu, principal investigator, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCvsT
Record Dates: First submitted 2012-01-29; First posted 2012-02-06 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Breast Cancer
Keywords: Metronomic cyclophosphamide; metastatic breast cancer; first line; docetaxel
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TC (Experimental): Docetaxel plus Cyclophosphamide
  Interventions: Drug: Docetaxel and Cyclophosphamide (TC)
- T (Active Comparator): Docetaxel
  Interventions: Drug: Docetaxel (T)

INTERVENTIONS:
Drug: Docetaxel and Cyclophosphamide (TC) — Docetaxel 75mg/m2 IVGTT D1 Cyclophosphamide 50mg PO D1-21;every 21days
  Arms: TC
Drug: Docetaxel (T) — Docetaxel 75mg/m2 IVGTT D1;every 21days
  Arms: T

SUMMARY:
The purpose of this study is to evaluate the role of metronomic cyclophosphamide in addition to docetaxel in first line therapy in metastatic breast cancer.

DETAILED DESCRIPTION:
Metronomic chemotherapy has been considered as an effective strategy for metastatic breast cancer. This trial is designed to evaluate the role of metronomic cyclophosphamide in addition to docetaxel in first line therapy in metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Females with age between 18 and 70 years old
2. ECOG performance between 0-1
3. Life expectancy more than 3 months
4. Histological proven unresectable recurrent or advanced breast cancer
5. No previous chemotherapy for metastatic breast cancer;suitable for monotherapy (Neoadjuvant or adjuvant docetaxel should be completed at least one year).
6. At least one measurable disease according to the response evaluation criteria in solid tumor (RECIST1.1)
7. No anticancer therapy within 4 weeks
8. Adequate hematologic, hepatic, and renal function,No serious medical history of heart, lung, liver and kidney
9. Provision of written informed consent prior to any study specific procedures

Exclusion Criteria:

1. Pregnant or lactating women (female patients of child-bearing potential must have a negative serum pregnancy test within 14 days of first day of drug dosing, or, if positive, a pregnancy ruled out by ultrasound)
2. Women of child-bearing potential, unwilling to use adequate contraceptive protection during the course of the study
3. Treatment with an investigational product within 4 weeks before the first treatment
4. Symptomatic central nervous system metastases
5. Other active malignancies (including other hematologic malignancies) or other malignancies, except for cured nonmelanoma skin cancer or cervical intraepithelial neoplasia.
6. Patient having a history of clinically significant cardiovascular, hepatic, respiratory or renal diseases, clinically significant hematological and endocrinal abnormalities, clinically significant neurological or psychiatric conditions
7. Uncontrolled serious infection
8. Patients with bad compliance

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 6 weeks

SECONDARY OUTCOMES:
Biomarker serum VEGF level | 6 weeks
  Relationship of serum VEGF level and efficacy
Biomarker immuno-marker | 6 weeks
  Relationship of immuno-marker(CD3,CD4,CD8 ect) and efficacy
Efficacy Overall Response Rate | 6 weeks
  Overall Response Rate
Efficacy Overall Survival | 6 weeks
  Overall Survival, OS
Safety | 6 weeks
  Safety（NCI CTCAE v4.0）
genetic polymorphisms | 6 weeks
  To evaluate the relationship of genetic polymorphisms and efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Zhonghua Wang, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China